CLINICAL TRIAL: NCT02911441
Title: Evaluating CBT Delivered by Community Health Workers on Maternal Mental Health and Infant Cognitive Development in Insecure Environments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heartland Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0721-03
Record Dates: First submitted 2016-09-19; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Maternal Anxiety; Maternal Depression; Infant Cognitive Development
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): Receives 8-12 weeks of one-on-one Cognitive Behavioral Therapy sessions
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Control Group (No Intervention): Receives no intervention during data-collection phase. Participants in this group will receive the intervention post-data collection.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy
  Arms: Treatment Group

SUMMARY:
This study evaluates a cognitive behavioral therapy intervention for mothers with symptoms of anxiety and depression living in insecure environments using a randomized controlled methodology. Key outcomes of interest include maternal mental health and infant cognitive development. The intervention will be delivered by community mental health workers who will be trained to administer 8 to 12 cognitive behavioral therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Women in their third trimester of pregnancy
* Who exhibited symptoms of anxiety and depression

Exclusion Criteria:

* Women who express suicidality

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Symptoms of anxiety and depression as measured by Hopkins Symptoms Checklist | 10 months post-birth of their infant
Infant Cognitive Development as measured by Mullen Scales of Early Learning | 10 months post-birth

CONTACTS AND LOCATIONS:
Overall Officials: Constantin Kahorha, Principal Investigator — Heartland Alliance International
Locations (1):
- Heartland Alliance International, Bukavu, South Kivu, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No